CLINICAL TRIAL: NCT05739175
Title: The Effect of Interactive Nurse Support Program Developed by Mobile Application on Patient Outcomes in Breast Cancer Patients Receiving Chemotherapy During the Coronavirus Pandemic.
Brief Title: The Effect of the Mobile Application-based Support Program on the Outcomes of Breast Cancer Patients in the Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, handan özdemir, Phd Candidate, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Zz123456.
Record Dates: First submitted 2022-07-07; First posted 2023-02-22 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Nursing
Keywords: Breast cancer; Nursing; Mobile Application; Pandemic; Symptom management
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group receiving interactive nurse support based on mobile application (Experimental): Experimental: Intervention Group The mobile application containing an interactive nurse support program will be uploaded to the telephone of the intervention group patients. Patients will be informed on how to use the mobile application. Data will be collected face-to-face before chemotherapy begins and by telephone one week after every four chemotherapy. Demographic/Clinical Information Form, Eastern Cooperative Oncology Group Performance Scale, Multidimensional scale of perceived social support, Memorial Symptom Rating Scale, European Organization for Research and Treatment of Cancer- Quality of Life, QLQ-BR23, Beck Anxiety Scale and Mobile Application evaluation form will be used to collect data.
  Interventions: Device: Mobile Application with Interactive Nurse Support
- Control group receiving standard care and no intervention (No Intervention): No Intervention: Control Group The patients received routine care and training in the polyclinic, and no additional intervention was applied. Data will be collected face-to-face before chemotherapy begins and by telephone one week after every four chemotherapy.Demographic/Clinical Information Form, Eastern Cooperative Oncology Group Performance Scale, Multidimensional scale of perceived social support, Memorial Symptom Rating Scale, European Organization for Research and Treatment of Cancer- Quality of Life, QLQ-BR23,Beck Anxiety will be used to collect data.

INTERVENTIONS:
Device: Mobile Application with Interactive Nurse Support — A mobile application containing an interactive nurse support program will be applied to the patients in the experimental group and its effect on patient outcomes will be evaluated through scales.
  The mobile application consists of three modules. The first part is a learning module with videos on Covid 19, breast cancer and chemotherapy related side effects management. Second part is ask the nurse/doctor. Third part is patient experiences module.
  After the participants download the mobile application to their phones, they can log in to the application with a valid e-mail address and password.
  Arms: Intervention group receiving interactive nurse support based on mobile application

SUMMARY:
Breast cancer remains the most common type of cancer in the world. Cancer itself and chemotherapy treatment, which is one of the most important treatment steps, may cause unwanted physical, social and psychological effects (symptoms) for the patient. These effects significantly affect the patient's quality of life. It is possible to manage the symptoms and reduce their destructive effects with professional care and treatment support that includes evidence-based practices. On the other hand, breast cancer patients receiving chemotherapy during the Coronavirus Pandemic form the risk group in terms of infection; On the one hand, the continued treatment and care support, on the other hand, required changes in the approach to the patient in order to reduce the risk of infection. In addition to reducing the risk of infection, mobile applications can create an alternative during the coronavirus Pandemic. process in order to maintain quality and uninterrupted care and treatment. This study is planned to be conducted analytically in a randomized controlled single-blind pattern in order to determine the effect of the interactive nurse support program developed with the mobile application on the patient outcomes (symptom management, quality of life, social support perception and anxiety) in breast cancer patients who received chemotherapy during the coronavirus pandemic. Within the scope of the study, interactive nurse support developed with mobile application will be applied to the research group from patients who apply to the polyclinic to receive chemotherapy treatment, and the control group will receive standard care. As a result of the analysis of the data collected systematically with forms and scales, the effect of the interactive nurse support program developed with the mobile application on patient outcomes (symptom management, quality of life, social support perception and anxiety) will be evaluated and recommendations will be made regarding the use of the application in patients with breast cancer.

DETAILED DESCRIPTION:
Type of Research:

This research is planned to be carried out as randomized controlled analytical in order to determine the effect of the interactive nurse support program developed with the mobile application in breast cancer patients receiving chemotherapy during the Coronavirus pandemic process.

Hypotheses of the Research:

H0-1: The interactive nurse support program developed with a mobile application in breast cancer patients receiving chemotherapy during the coronavirus pandemic is not effective on patients' perception of social support.

H0-2: The interactive nurse support program developed with a mobile application in breast cancer patients receiving chemotherapy during the coronavirus pandemic. process is not effective on symptom management (symptom frequency, severity, level of distress).

H0-3: The interactive nurse support program developed with a mobile application in breast cancer patients receiving chemotherapy during the coronavirus pandemic. is not effective on the quality of life of the patients.

H0-4: The interactive nurse support program developed with a mobile application in breast cancer patients receiving chemotherapy during the coronavirus pandemic is not effective on patients' anxiety levels.

Population and Sample of the Research:

The population of the study consists of all breast cancer patients who applied to Ankara City Hospital Medical Oncology Department Outpatient Clinic to receive chemotherapy treatment.

In order to determine the sample size, a similar study (Zhu et al. 2018) was examined, and since the measurement tools were different, this study could not be used in calculating the sample number. However, when similar studies using mobile applications were examined in terms of sample size, it was seen that the number of patients in the intervention and control groups was 50 or less. For this reason, first of all, after the twelve-week follow-up of 50 patients in the control group is completed, the mobile application will be applied to 10 patients from the intervention group. When the twelve-week follow-up of 10 patients from the intervention group is completed, a power analysis will be made with the G. Power program using the data of 10 patients in each group, and the minimum number of people to be sampled will be calculated. The number of patients in the control group and intervention group will be increased according to the minimum number of people calculated. In order to prevent possible interaction between the patients, data will be collected from the intervention group patients after the follow-up of the control group patients is completed

Randomization Method:

During the preliminary implementation of the study, it was learned that based on the new working procedure of the Outpatient Chemotherapy Unit, all breast cancer patients who received anthracycline-based chemotherapy were given a treatment appointment at the same time in the afternoon. It was also found that the patients received chemotherapy in the same time interval in side-by-side seats and that the risk of mutual interaction was quite high. Contamination because of interaction between the intervention and control groups causes potential bias in the evaluation of the effect of the intervention in randomized controlled experimental studies. For this reason, patients who met the inclusion criteria were assigned to the intervention and control groups in a way that they would not come into contact with each other. To this end, the Simple Randomization Technique was used to determine which group the data would be collected from first (Random.org, 2021). Since the first group was determined as the control group in the randomization, the data were collected from this group first and then from the intervention group.

Data Collection Tools:

1. Demographic and Clinical Information Form
2. ECOG (Eastern Cooperative Oncology Group) Performance Scale
3. Multidimensional Scale of Perceived Social Support (MSPSS)
4. Memorial Symptom Rating Scale (MSDS)
5. European Organization for Research and Treatment of Cancer- Quality of Life (EORTC-QLQ) C30 Scale
6. QLQ-BR23 Module
7. Beck Anxiety Scale
8. Mobile Application Effectiveness Evaluation Form Pre-application In order to evaluate the comprehensibility and usability of the mobile application and data collection forms created for the interactive nurse support program, a preliminary application was made with 5 patients who met the criteria for inclusion in the study among the patients who applied to the Ankara City Hospital Medical Oncology Department Outpatient Clinic with the diagnosis of Breast Cancer to receive chemotherapy treatment. will be done. After the preliminary application, necessary changes will be made in the mobile application and data collection forms. If changes are made in the mobile applications and forms in line with the pre-application, the patients included in the pre-application will not be included in the research sample

Application of the Research:

Part 1: Development of Mobile Application 1.1.Developing the Content of the Mobile Application The content of the mobile application will be created by the researcher as a result of extensive literature research. The content created will be submitted to expert opinion, including 1 oncologist, 1 surgical oncology specialist, 4 nurse lecturers, 1 Turkish Linguist, 1 psychiatrist, 1 psychologist and 2 oncology nurses. At the same time, the content of the mobile application will be examined by 3 breast cancer patients and its intelligibility will be evaluated. As a result of expert opinions and patient evaluations, arrangements will be made in the content of the mobile application and the mobile application will be finalized.

The mobile application content will consist of 5 parts:

1. Coronavirus Pandemic Information Module
2. Learning Module
3. Discussion Module
4. Ask the Expert Module
5. Lived Stories Module 1.2. Creating the Technical Infrastructure of the Mobile Application The technical infrastructure of the application will be developed by the web software engineer.

Part 2: Implementation of Mobile Application and Collection of Data

* Patients with breast cancer who apply to the Department of Medical Oncology will be identified.
* Patients with breast cancer who meet the inclusion criteria will be identified (ECOG Performance Scale will be applied at this stage )
* Oral and written information will be given to the patients who are planned to be included in the study at the beginning of the study, and Informed Voluntary Consent Forms will be filled and signed according to their acceptance status.
* The first day of chemotherapy for patients who meet the inclusion criteria and accept to participate in the study will be determined. An appointment will be made one day before the chemotherapy treatment and data collection forms will be applied (day 0).

Practices for Patients in the Intervention Group

* Interviewing the patients in the intervention group the day before chemotherapy starts (day 0); *Demographic and Clinical Information Form

  * Multidimensional Scale of Perceived Social Support
  * EORTC QLQ-C30 Quality of Life Scale and QLQ-BR23 Module
  * Beck Anxiety Scale will be applied.
* The mobile application will be installed on the patient's phone by the researcher. The patient will be registered to the program by creating a changeable user name.
* The patient will be given 15-20 minutes of training on the use of the mobile application.
* The mobile application will be applied during 4 cycles of chemotherapy (1 cycle/3 weeks or 1 cycle/2 weeks) from the first day of chemotherapy treatment.

The patient will record the symptoms (symptom type and severity) on the mobile application since the first chemotherapy treatment, and watch the relevant video recording according to the symptom experienced from the symptom management videos. The patient will be informed that he can record more than one symptom and watch all the videos as many times as he wants. Information texts on patient breast cancer and coronavirus will also be accessible at all times. This section covers the "Learning Module" of the mobile application.

* In addition to the video recording, which includes the management initiatives for the symptom experienced by the patient, the patient will forward his/her individual questions to the researcher by text message or phone call, according to his/her preference. According to the method of conveying the patient's question, the patient's question will be answered by the researcher with the same method. As soon as written messages are sent, they will appear on the researcher's phone screen and the patient will be answered within 1 hour at the latest. If necessary according to the content of the questions regarding the treatment, care or symptom management submitted by the patient, the questions will be directed to the oncology physician, who is the other manager in the Ask the Specialist module. The response from the physician will be communicated to the patient. This section covers the "Ask an Expert Module" of the mobile application.
* A reminder message will be sent to the patients who do not register their symptoms and log in to the system during the day, as of 20:00.

Patients will be able to enter the Discussion Module according to their preferences and share their experiences and opinions with other patients in the research group who have had the same experiences. This section covers the "Discussion Module" of the mobile application.

* Patients will be able to watch video recordings containing interviews with patients who have had the same experience and have come to the end of their treatment, whenever they want and as many times as they want. This section covers the "Lived Stories Module" of the mobile application.
* Patients will use the mobile application for 8 weeks or 12 weeks after receiving the first course of chemotherapy. Data will be collected with Multidimensional Perceived Social Support Scale, Memorial Symptom Rating Scale, EORTC QLQ-C30 Quality of Life Scale, QLQ-BR23 Module, Beck Anxiety Scale before chemotherapy is started and after each chemotherapy course, 4 times in total. When the cures are completed, a Mobile Application Efficiency Evaluation Form will be added to the data collection forms.

Applications for the Patients in the Control Group:

* The mobile application will not be installed on the phones of the patients in the control group, and the patients will receive standard care.
* Standard care; It includes the patients receiving chemotherapy in the outpatient clinic during the cure times given to them and informing the chemotherapy nurse about the pre-chemotherapy process and possible symptoms.
* Control group patients will be followed for 8 weeks or 12 weeks (4 cycles). Data will be collected with Multidimensional Perceived Social Support Scale, Memorial Symptom Rating Scale, EORTC QLQ-C30 Quality of Life Scale, QLQ-BR23 Module, Beck Anxiety Scale, before chemotherapy starts and after each chemotherapy cycle, 4 times in total.

Dependent and Independent Variables of the Research; Dependent Variables of the Research; symptom management, quality of life, perception of social support, level of anxiety. The independent variables of the research; sociodemographic and clinical characteristics of the patient, interactive nurse support mobile application Evaluation of Data The data to be obtained from the research will be analyzed with the SPSS 22 Program. Descriptive statistics (number, percentage, mean) will be used in the evaluation of the data. The relationship between the measured variables will be evaluated with the t-test, Pearson Chi-square test and Fishher's exact test. In the analysis of multiple dependent variables, 2-way Analysis of Variance and Regression Analysis will be used. A value of p<0.05 will indicate that the difference is significant, and a value of p>0.05 will indicate that the difference is not significant.

Ethical Dimension of Research Necessary permissions will be obtained from Ankara City Hospital in order to carry out the research. Written consent will be obtained from the patients to be included in the study with Informed Consent Forms.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Volunteering to participate in the research,
* Having been diagnosed with breast cancer (Stage 0,1,2),
* Being able to understand and speak Turkish,
* ECOG performance scale score of 0, 1 and 2
* Being literate
* Owning a mobile phone with Android or iphone operating system processor and using the phone effectively
* Receiving chemotherapy treatment for the first time

Exclusion Criteria:

* Refusal to participate in the research,
* Diagnosing metastatic breast cancer (Stage 3,4),
* Receiving simultaneous radiotherapy or biotherapy with chemotherapy,
* Having visual, auditory or mental problems,
* Having a psychiatric diagnosis,
* Those who have received chemotherapy before
* ECOG performance scale score of 3 and 4,
* Taking part in another research that will affect the research results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 100 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Change of EORTC QLQ-C30 Quality of Life Scale and QLQ-BR23 Module score at baseline and one week later after first, second, third and fourth chemotherapy. | The first measurement will be made before chemotherapy. The second, third, fourth, and fifth measurement will be made one week after the first, second, third, and fourth chemotherapy, respectively.
  EORTC QLQ-C30 Quality of Life Scale was developed by Aronson in 1993.Turkish validity and reliability of the scale made by Beşer and Öz in 2003.The scale consists of three subgroups as general well-being, functional area and symptoms and includes 30 questions for the past week. The first 28 of the 30 items in the scale are a four-point Likert scale. In the 29th question of the scale, the patient is asked to evaluate his health on a scale of 1 to 7 (1: very poor and 7: excellent), and in the 30th question, the general quality of life.High functional area and general well-being subgroup scores and low symptom subgroup scores indicate a high quality of life. EORTC QLQ-BR23 Breast Cancer Module was developed by Srangers at al. in 1996.It consists of 23 items.High functional dimension scores indicate high quality of life. A high score on the symptoms dimension indicates a low quality of life.
Change of Memorial Symptom Assesment Scale score at baseline and one week later after first, second, third and fourth chemotherapy. | The first measurement will be made before chemotherapy. The second, third, fourth, and fifth measurement will be made one week after the first, second, third, and fourth chemotherapy, respectively.
  Memorial Symptom Assesment Scale was developed by Portenoy et al. in 1994. Turkish validity and reliability of the scale made by Yıldırım et al. in 2011. The scale is used to evaluate the frequency and severity of symptoms experienced by cancer patients during the past seven days. It consists of 32 symptoms. While the 'frequency' and 'intensity' levels of the symptoms are answered as a 4-point likert, the 'distress' levels are answered as a 5-point likert. Total score is obtained by averaging thirty-two symptom scores. Each symptom score is calculated by averaging the frequency, severity, and degree of distress.
Change of Multidimensional Scale of Perceived Social Support score at baseline and one week later after first, second, third and fourth chemotherapy. | The first measurement will be made before chemotherapy. The second, third, fourth, and fifth measurement will be made one week after the first, second, third, and fourth chemotherapy, respectively.
  Multidimensional Scale of Perceived Social Support was developed by Zimet et al. in 1988. Turkish validity and reliability of MSPSS was performed by Eker et al. MSPSS consists of 12 items and 3 sub-dimensions that subjectively evaluate the adequacy of social support from three different sources. These sub-dimensions are family, friends, and a special person. Each item was rated using a 7-point scale. The person to whom the scale was applied can give at least 1 point to the sentence that he disagreed with, and maximum 7 points to the sentence that he agrees with. As the score given to each item increases, the perceived social support also increases. Any score between 12 and 84 (min.-max.) can be obtained from the scale. The Cronbach Alpha coefficient of the scale is 0.89
Change of Beck Anxiety Inventory scale score at baseline and one week later after first, second, third and fourth chemotherapy. | The first measurement will be made before chemotherapy. The second, third, fourth, and fifth measurement will be made one week after the first, second, third, and fourth chemotherapy, respectively.
  Beck Anxiety Scale was developed by Aeron T. Beck in 1988 to measure anxiety in cancer It was translated into Turkish by Ulusoy et al in 1998 and validated. İtems in the scale describe the subjective, somatic and panic symptoms of anxiety. The scores obtained from all items are summed as "0=none, 1=mild, 2=moderate, 3=severe" for each item. The score range is between 0-63 (min.-max.) 8-15 points indicates mild anxiety, 16-25 points indicates moderate anxiety, 26-63 points indicates severe anxiety. A high total scale score indicates high anxiety. The Cronbach Alpha coefficient of the scale is 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Doğan Uncu, professor, Study Director — Ankara Bilkent Central Hospital
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozdemir H, Demir A, Bardakci M, Uncu D. The effect of an interactive nurse support program developed with a mobile application on patient outcomes in breast cancer patients who received outpatient chemotherapy: A randomized controlled trial. Eur J Oncol Nurs. 2025 Jun;76:102882. doi: 10.1016/j.ejon.2025.102882. Epub 2025 Mar 25. PMID 40185060